CLINICAL TRIAL: NCT01928979
Title: Retrospective Registry Providing Baseline Data on the Outcome of Left Atrial (LA) or LA Appendage (LAA) Thrombus in Patients With Nonvalvular Atrial Fibrillation (AF) or Atrial Flutter After Standard of Care (SoC) Anticoagulant Therapy
Acronym: CLOT-AF
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16677; NN1301 (Other: company internal)
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: LA/LAA Thrombus; Atrial Fibrillation; Observation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: no drug

INTERVENTIONS:
Other: no drug — Patients who suffered from hemodynamically stable nonvalvular AF or atrial flutter and had a diagnosed LA/ LAA thrombus between January 1st, 2011 and December 31st, 2012

SUMMARY:
Thrombus outcome data will be collected retrospectively during 2011-2012 as a historical baseline of SoC with oral VKA (Vitamin K Antagonist(s) for the treatment of patients with nonvalvular AF or atrial flutter documented with LA/ LAA thrombi on transesophag-eal echocardiography (TEE).

The study is a company-sponsored, global, multi-center, retrospective, non-interventional study. Patients who suffered from hemodynamically stable nonvalvular AF or atrial flutter and had a diagnosed LA/ LAA thrombus between January 1st, 2011 and December 31st, 2012 will be identified through screening and review of medical records and included in the registry. Retrospective patient data will be collected from May 2nd, 2013 to May 2nd, 2014. The observation of each patient will cover the period from the diagnosis of an LA/ LAA thrombus until the end-of-treatment TEE following the 3-12 week SoC anticoagulation (AC) therapy. If no end-of-treatment TEE has been performed during 3-12 weeks of AC therapy, the observational period will end at 12 weeks after diagnosis at the latest. If more than one TEE was performed during treatment, the thrombus outcome will be collected from the last TEE performed within 12 weeks of treatment start.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age ≥ 18 years at data recording
* Hemodynamically stable nonvalvular AF or atrial flutter
* Documented LA/ LA thrombus on TEE

Exclusion Criteria:

* Valvular AF ( ESC 2012 definition)
* History of cardiac thrombus confirmed on TEE
* Intracardiac tumors, e.g. atrial myxoma
* Active endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who suffered from hemodynamically stable nonvalvular AF or atrial flutter and had a diagnosed LA/ LAA thrombus between January 1st, 2011 and December 31st, 2012.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2013-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Thrombus resolution (completely disappeared) rate confirmed on TEE. | after 3-12 weeks of SoC treatment or lost to follow up, whichever is later

SECONDARY OUTCOMES:
Stroke or non central nervous system (CNS) systemic thromboembolism rate | after 3-12 weeks of SoC treatment or lost to follow up, whichever is later
All bleeding (major, non-major, unknown severity) rates | after 3-12 weeks of SoC treatment or lost to follow up, whichever is later

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Many Locations, Bulgaria
- Many Locations, France
- Many Locations, North Rhine-Westphalia, Germany
- Many Locations, Poland
- Many Locations, Russia
- Many Locations, Turkey (Türkiye)
- Many Locations, Ukraine

REFERENCES:
- [Derived] Lip GY, Hammerstingl C, Marin F, Cappato R, Meng IL, Kirsch B, Morandi E, van Eickels M, Cohen A. Rationale and design of a study exploring the efficacy of once-daily oral rivaroxaban (X-TRA) on the outcome of left atrial/left atrial appendage thrombus in nonvalvular atrial fibrillation or atrial flutter and a retrospective observational registry providing baseline data (CLOT-AF). Am Heart J. 2015 Apr;169(4):464-71.e2. doi: 10.1016/j.ahj.2014.12.020. Epub 2015 Jan 6. PMID 25819852